CLINICAL TRIAL: NCT04797715
Title: A Double-blind, Placebo-controlled, Randomized Withdrawal Trial to Assess the Efficacy and Safety of AXS-05 for the Treatment of Agitation in Subjects With Dementia of the Alzheimer's Type
Brief Title: Assessing Clinical Outcomes in Alzheimer's Disease Agitation
Acronym: ACCORD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-05-AD-302
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type; Alzheimer Disease; Agitation,Psychomotor
Keywords: AD agitation; AXS-05; NMDA receptor antagonist; dextromethorphan; bupropion; Axsome; ACCORD
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (Experimental): Up to 26 weeks in double-blind period
  Interventions: Drug: AXS-05
- Placebo (Placebo Comparator): Up to 26 weeks in double-blind period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 — AXS-05 tablets, taken twice daily
  Arms: AXS-05
Drug: Placebo — Placebo tablets, taken twice daily
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, placebo-controlled, randomized withdrawal study to evaluate the efficacy and safety of AXS-05 compared to placebo in the treatment of agitation symptoms in subjects with agitation associated with Alzheimer's disease.

DETAILED DESCRIPTION:
Enrolled patients will first enter a 9-week, open-label stabilization period, during which they will be treated with AXS-05 and monitored for a treatment response. Patients who experience a treatment response during the stabilization period will then be randomized into the double-blind treatment period, in a 1:1 ratio, to continue treatment with AXS-05 or to switch to placebo, for up to 26 weeks or until a relapse of agitation occurs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) based on the 2011 National Institute on Aging-Alzheimer Association (NIA-AA) criteria.
* Diagnosis of clinically signification agitation resulting from probable AD according to the International Psychogeriatric Association (IPA) provisional definition of agitation.

Exclusion Criteria:

* Patient has dementia predominantly of non-Alzheimer's type.
* Patient has symptoms of agitation that are not secondary to AD (e.g., pain, other psychiatric disorder or delirium due to a metabolic disorder, systemic infection, or substance-induced).
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Time from randomization to relapse of agitation symptoms | up to 26 weeks

OTHER OUTCOMES:
Types and rates of adverse events | up to 35 weeks

CONTACTS AND LOCATIONS:
Locations (60):
- United States (58):
  - Clinical Research Site, Sun City, Arizona
  - Clinical Research Site, Tucson, Arizona
  - Clinical Research Site, Chula Vista, California
  - Clinical Research Site, Imperial, California
  - Clinical Research Site, Lafayette, California
  - Clinical Research Site, Los Alamitos, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Temecula, California
  - Clinical Research Site, Coral Springs, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, Lake City, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Naples, Florida
  - Clinical Research Site, Ocoee, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Pembroke Pines, Florida
  - Clinical Research Site, Pensacola, Florida
  - Clinical Research Site, St. Petersburg, Florida
  - Clinical Research Site, Sunrise, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Trinity, Florida
  - Clinical Research Site, Augusta, Georgia
  - Clinical Research Site, Columbus, Georgia
  - Clinical Research Site, Suwanee, Georgia
  - Clinical Research Site, Honolulu, Hawaii
  - Clinical Research Site, Boise, Idaho
  - Clinical Research Site, Wichita, Kansas
  - Clinical Research Site, Bangor, Maine
  - Clinical Research Site, Lowell, Massachusetts
  - Clinical Research Site, Flint, Michigan
  - Clinical Research Site, Chesterfield, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, East Syracuse, New York
  - Clinical Research Site, New Windsor, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Charlotte, North Carolina
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Dayton, Ohio
  - Clinical Research Site, Jenkintown, Pennsylvania
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Cypress, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, McKinney, Texas
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Sugar Land, Texas
  - Clinical Research Site, West Jordan, Utah
  - Clinical Research Site, Woodstock, Vermont
  - Clinical Research Site, Everett, Washington
  - Clinical Research Site, Waukesha, Wisconsin
- Canada (2):
  - Clinical Research Site, Kelowna, British Columbia
  - Clinical Research Site, Newmarket, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://axsome.com/